## **Study Title**

Effect of Arthroscopic Microfracture Combined with Stromal Vascular Fraction Therapy on Clinical and Radiological Outcomes in Gonarthrosis: A Prospective Randomized Controlled Trial

### **NCT Number**

NCT07112885

# Organization

Istanbul University, Department of Orthopedics and Traumatology

### **Document Date**

**September** 19, 2025

## Informed Consent Form

StudyTitle: ComparisonofSVF InjectionWith andWithout Microfracture in Moderate Knee

Osteoarthritis

Institution: Istanbul University, Department of Orthopedics and Traumatology

#### Introduction

You are invited to participate in a clinical study investigating the effects of stromal vascular fraction (SVF) injection with and without microfracture in patients with moderate knee osteoarthritis. Before you decide, it is important that you understand the purpose of the study, what it involves, and any possible risks or benefits.

## Purpose of the Study

The purpose of this study is to compare the clinical and radiological outcomes of two different treatment methods in patients with moderate knee osteoarthritis: (1) arthroscopic debridement and microfracture followed by intra-articular SVF injection, and (2) arthroscopic debridement followed by SVF injection alone.

#### **Procedures**

If you agree to participate, you will be randomly assigned to one of two groups. All patients will undergo arthroscopic knee debridement. Group A will receive additional microfracture and SVF injection, while Group B will receive SVF injection alone. Follow-up visits will be conducted at baseline, 3, 6, 12, and 24 months, with MRI imaging performed at baseline, 12, and 24 months.

#### **Risks and Discomforts**

Possible risks include pain, swelling, stiffness, or infection after the procedure. As with any surgical or injection procedure, there is a small risk of complications related to anesthesia or the intervention itself.

#### **Benefits**

Potential benefits may include reduced pain, improved knee function, and possible improvement in cartilage quality. However, there is no guarantee of direct personal benefit.

## Confidentiality

All information collected during the study will be kept strictly confidential. Your identity will not be disclosed in any publication or report.

## **Voluntary Participation**

Participation in this study is entirely voluntary. You may refuse to participate or withdraw at any time without giving a reason, and this will not affect your standard medical care.

#### **Contact Information**

If you have any questions or concerns about the study, please contact the principal investigator: Dr. Mehmet Yağız Yenigün Istanbul University, Department of Orthopedics and Traumatology

### Consent

I have read and understood the information provided above. I voluntarily agree to participate in this study.

| Participant Name and Signature: |
|---------------------------------|
| Oate: |
| nvestigator Name and Signature: |

### **Ethical Considerations**

The study protocol was approved by the Institutional Review Board of Istanbul University. All patients provided written informed consent prior to participation.



**Ethics Approval-English Version** 

**Reference:** Letter of the Department of Orthopedics and Traumatology dated 06/04/2022 and numbered 839487

The study titled "Comparison of the Clinical and Radiological Outcomes of Isolated Intra-articular SVF (Stromal Vascular Fraction–Stem Cell) Therapy with Arthroscopic Microfracture (Debridement) + SVF Therapy", with file number 2023/106, for which you are the principal investigator and conducted by Dr. Mehmet Yağız YENİGÜN, was reviewed at the meeting of our committee dated 20/01/2023 and numbered 02, and it was found to be ethically appropriate. The minutes of the meeting are attached.

For your information.

**Document Verification Code: BSNV6R250P** 

**PIN Code: 42152** 

Prof. Dr. Ali Yağız ÜRESİN Chairman of the Committee

#### Note:

Asubsequent ethics committee application was submitted in order to increase the number of participants (from 40 to 50) and to update the study title. This amendment request was reviewed and approved by the committee, confirming that both the protocol modification and the revised sample size were ethically appropriate.



Ethics Approval-English Version

**Reference:** Letter of the Department of Orthopedics and Traumatology dated 17/03/2025 and numbered 3241799

The study titled "Comparison of the Clinical and Radiological Outcomes of Isolated Intra-articular SVF (Stromal Vascular Fraction–Stem Cell) Therapy with Arthroscopic Microfracture (Debridement) + SVF Therapy", with file number 2023/106, for which you are the principal investigator and conducted by Dr. Mehmet Yağız YENİGÜN, was reviewed at the meeting of our committee dated 20/01/2023 and numbered 02, and was found to be ethically appropriate.

Your request for amendment, including the Amendment Information Form, the change in the number of participants (from 40 to 50), and the thesis title modification from "Comparison of the Clinical Outcomes of Isolated Intra-articular SVF Therapy with Arthroscopic Debridement + SVF Therapy" to "Effect of Arthroscopic Microfracture Combined with Stromal Vascular Fraction Therapy on Clinical and Radiological Outcomes in Gonarthrosis: A Prospective Randomized Controlled Trial", was reconsidered at the meeting of our committee dated 18/04/2025 and numbered 08, and was also found ethically appropriate. The minutes of the meeting are attached.

For your information.

**Document Verification Code: BS93BP48J8C** 

**PIN Code: 26213** 

Prof. Dr. Ali Yağız ÜRESİN Chairman of the Committee